CLINICAL TRIAL: NCT04191681
Title: Safety and Efficacy of Angiotensin Receptor-neprilysin Inhibitor After Left Ventricular Assist Device ImplanT (SEAL-IT) Study
Brief Title: Safety and Efficacy of ARNI After LVAD ImplanT (SEAL-IT) Study
Acronym: SEAL-IT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Jerry Estep MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-1132
Record Dates: First submitted 2019-11-18; First posted 2019-12-10 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Stage D Heart Failure
Keywords: continuous flow left ventricular assist device; sacubitril-valsartan; oral vasodilator; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Standard of Care; Vasodilator Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril-valsartan study arm (Experimental): 1. Start medication-naïve patients on low-dose sacubitril-valsartan (24/26 mg PO BID) without a washout period per guideline and label recommendations.
  2. Switch patients to equivalent dose sacubitril-valsartan if on prior ACE inhibitor (after a 36 hour washout period) or ARB therapy (after discontinuing one day prior).
  3. If therapeutic range MAP (65 to 85 mm Hg), discontinue other oral vasodilator (e.g., hydralazine, isordil) or non-rate limiting dihydropyridine calcium channel blocker (non-DHP CCB, e.g., amlodipine) therapy on the day prior to sacubitril-valsartan initiation. If MAP > 85 mm Hg, low-dose sacubitril-valsartan will be added with or without discontinuation of other oral vasodilator or non-DHP CCB per physician's discretion based on drug tolerability and maintenance of therapeutic range MAP.
  4. Sacubitril-valsartan can be up-titrated every 2-4 weeks per standard practice guidelines per physician's discretion as above.
  Interventions: Drug: Sacubitril-Valsartan
- Usual care (standard-of-care) arm (Active Comparator): 1. Continue current regimen of patients on oral vasodilator therapy (e.g., ACE inhibitor, ARB, hydralazine, isordil), allowing for up-titration of the drug every 2-4 weeks per standard practice guidelines in keeping with physician's discretion as above.
  2. Start medication-naïve patients de novo on one of the oral vasodilators as below per guideline and label recommendations, allowing for up-titration of the drug every 2-4 weeks per standard practice guidelines in keeping with physician's discretion as above: i. ACE inhibitor: Enalapril 2.5 mg PO BID or Lisinopril 5 mg PO daily; ii. ARB: Valsartan 20 mg PO BID or Losartan 25 mg PO daily; iii. Other: Hydralazine 10 mg PO TID or Isordil 5 mg PO TID.
  Interventions: Drug: Usual care (standard-of-care) arm

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Sacubitril-valsartan at low or equivalent dose to be initiated or added to patients randomized to this arm, and titrated up every 2-4 weeks, per standard practice guidelines and label recommendations per physician's discretion.
  Other Names: Entresto
  Arms: Sacubitril-valsartan study arm
Drug: Usual care (standard-of-care) arm — Other oral vasodilator therapy to be continued or initiated to patients randomized to this arm, and titrated up every 2-4 weeks, per standard practice guidelines and label recommendations per physician's discretion.
  Other Names: Oral Vasodilator
  Arms: Usual care (standard-of-care) arm

SUMMARY:
The purpose of the study is to evaluate how well tolerated and effective an angiotensin receptor-neprilysin inhibitor (sacubitril-valsartan) is in patients with contemporary durable continuous flow left ventricular assist device (CF-LVAD) implantation compared to usual care oral vasodilator therapy.

DETAILED DESCRIPTION:
The aim of this pilot study is to prospectively determine the short-term (at 3 months) and long-term (at 6 and 12 months) safety and efficacy of an angiotensin receptor-neprilysin inhibitor (sacubitril-valsartan) in patients with contemporary durable continuous flow left ventricular assist device (CF-LVAD) implantation compared to standard-of-care (usual care) oral vasodilator therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18 years)
2. Durable CF-LVAD for any indication
3. NYHA II to IV classification
4. LVEF < 40%
5. Written informed consent

Exclusion Criteria:

1. Inability to comply with the conditions of the protocol
2. Any patient with durable CF-LVAD who has any one of the following:

   i. symptomatic hypotension or MAP < 60 mm Hg at randomization,

   ii. eGFR < 30 mL/min/1.73 m2 at randomization,

   iii. potassium > 5.4 mM at randomization,

   iv. history of angioedema at randomization,

   v. history of unacceptable side effects with ACE inhibitor, ARB, or sacubitril-valsartan therapy at randomization,

   vi. use of vasoactive agents (e.g., dobutamine, dopamine, epinephrine, norepinephrine, phenylephrine, vasopressin, nitroglycerin, nitroprusside, epoprostenol) or parenteral diuretics in 24 hours preceding randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of drug discontinuation from drug-related adverse events due to sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 3 months | 3 months
  Incidence of drug discontinuation from drug-related adverse events due to sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 3 months. Incidence of drug discontinuation is defined as the number of patients exposed to the drug with an adverse event over the total number of patients exposed to the drug. An adverse event is defined as any one of the following: acute kidney injury with eGFR decline > 25% from baseline, hyperkalemia with potassium > 5.5 mM, hypotension with mean arterial pressure (MAP) < 60 mm Hg, angioedema, dizziness, and/or cough.
Time-averaged proportional change in NT-proBNP concentration (pg/mL) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 3 months | 3 months
  Time-averaged proportional change in NT-proBNP concentration (pg/mL) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 3 months.

SECONDARY OUTCOMES:
Time-averaged proportional change in NT-proBNP concentration (pg/mL) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 and 12 months | 6 and 12 months
  Time-averaged proportional change in NT-proBNP concentration (pg/mL) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 and 12 months.
Proportion of patients (%) with effective MAP control (65 to 85 mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 3, 6 and 12 months | 3, 6 and 12 months
  Proportion of patients (%) with effective MAP control (65 to 85 mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 3, 6 and 12 months.
Proportion of patients (%) on other cardiac medications with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 3, 6 and 12 months relative to baseline | 3, 6 and 12 months
  Proportion of patients (%) on other cardiac medications (e.g., diuretics, aldosterone antagonists, beta-blockers, oral vasodilators, and anti-hypertensives) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 3, 6 and 12 months relative to baseline.
Proportion of patients (%) in each New York Heart Association (NYHA) classification with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 3, 6 and 12 months relative to baseline | 3, 6 and 12 months
  Proportion of patients (%) in each New York Heart Association (NYHA) classification (e.g., functional class I-IV) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 3, 6 and 12 months relative to baseline.
Proportion of patients (%) with heart failure readmissions with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 and 12 months | 6 and 12 months
  Proportion of patients (%) with heart failure readmissions with sacubitril-valsartan versus standard-of-care oral vasodilator therapy determined at 6 and 12 months.
Absolute change in mean left ventricular end-diastolic dimension (mm) on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in mean left ventricular end-diastolic dimension (mm) on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in mitral E/A ratio on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in mitral E/A ratio on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in indexed left atrial volume (mL/m2) on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in indexed left atrial volume (mL/m2) on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in indexed right atrial volume (mL/m2) on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in indexed right atrial volume (mL/m2) on echocardiogram with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in mean right atrial pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in mean right atrial pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in mean pulmonary artery pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in mean pulmonary artery pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in mean pulmonary artery diastolic pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in mean pulmonary artery diastolic pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in mean pulmonary capillary wedge pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in mean pulmonary capillary wedge pressure (mm Hg) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in pulmonary artery pulsatility index with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in pulmonary artery pulsatility index with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in pulmonary vascular resistance (Woods Unit) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in pulmonary vascular resistance (Woods Unit) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in systemic vascular resistance (dynes-sec/cm5) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in systemic vascular resistance (dynes-sec/cm5) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.
Absolute change in cardiac index (L/min/m2) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy at 6 weeks and/or 3, 6 and/or 12 months | 6 weeks and/or 3, 6 and/or 12 months
  Absolute change in cardiac index (L/min/m2) with sacubitril-valsartan versus standard-of-care oral vasodilator therapy evaluated at 6 weeks and/or 3, 6 and/or 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry D Estep, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Duffy CI, Ambrosy AP, McCague K, Rocha R, Braunwald E; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Acute Decompensated Heart Failure. N Engl J Med. 2019 Feb 7;380(6):539-548. doi: 10.1056/NEJMoa1812851. Epub 2018 Nov 11. PMID 30415601
- [Background] Wachter R, Senni M, Belohlavek J, Straburzynska-Migaj E, Witte KK, Kobalava Z, Fonseca C, Goncalvesova E, Cavusoglu Y, Fernandez A, Chaaban S, Bohmer E, Pouleur AC, Mueller C, Tribouilloy C, Lonn E, A L Buraiki J, Gniot J, Mozheiko M, Lelonek M, Noe A, Schwende H, Bao W, Butylin D, Pascual-Figal D; TRANSITION Investigators. Initiation of sacubitril/valsartan in haemodynamically stabilised heart failure patients in hospital or early after discharge: primary results of the randomised TRANSITION study. Eur J Heart Fail. 2019 Aug;21(8):998-1007. doi: 10.1002/ejhf.1498. Epub 2019 May 27. PMID 31134724